CLINICAL TRIAL: NCT03412825
Title: The Effect of Dietary Supplementation on Nutrient Status in Families Living in a Food Insecure Environment
Brief Title: Diet, Nutrient Status, and Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 70573
Record Dates: First submitted 2018-01-08; First posted 2018-01-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Food Insecurity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Supplementation (Experimental)
  Interventions: Dietary Supplement: Egg supplementation
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Egg supplementation — Participants will required to consume 2 eggs per day, 5 days a week (a total of 10 eggs per week).
  Arms: Nutrition Supplementation

SUMMARY:
Arkansas has one of the highest rates for food insecurity and 27.7% of children in the University of Arkansas area are food insecure. In addition, more than 14% of children ages 2-4 are obese and 20% of children ages 10-17 are obese. In Northwest Arkansas, the area surrounding the University of Arkansas in Fayetteville (Washington County), the food insecurity rate for adults is 17.9% (an estimated 34,730 individuals) and the food insecurity rate for children under 17 years of age is 24.4% (12,150 individuals). In addition, the surrounding counties have similar food insecurity rates (This makes Northwest Arkansas an ideal location to conduct a pilot study focusing on egg supplementation, childhood obesity, and food insecurity (http://www.feedingamerica.org/hunger-in-america/our-research/map-the-meal-gap).

ELIGIBILITY:
Inclusion Criteria:

* Food insecurity assessed by use of SNAP benefits or qualifying using the US Food Security Scale).

Exclusion Criteria:

* No dietary restrictions
* Fear of needles
* Metabolic disorders
* Picky eating
* Taking medication

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Micronutrient status in plasma | The change in micronutrient status (e.g. iron, vitamin A, vitamin B12) will be measured from baseline to 16 weeks to determine if the dietary intervention improves baseline micronutrient status.
  Micronutrients status will be measured using plasma samples.
Body composition | The change in body composition (e.g. ratio of lean to fat mass) will measured from baseline to 16 weeks.
  Body composition will be measured using dual X-ray absorptiometry (DEXA) .

SECONDARY OUTCOMES:
Height | The change in height will be measured from baseline to 16 weeks.
  Height (in centimeters) will be measured using a stadiometer.
Weight | The change in weight will be measured from baseline to 16 weeks.
  Weight (in kilograms) will be measured using a scale.
Waist-to-hip ratio | The change in waist-to-hip ratio will be measured from baseline to 16 weeks.
  Waist-to-hip ratio will be measured using the protocol outlined by the World Health Organization.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie I Baum, PhD, Principal Investigator — University of Arkansas, Fayetteville
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No